CLINICAL TRIAL: NCT06546722
Title: Transversus Thoracic Plane Block for Perioperative Analgesia in Cardiac Surgery: a Randomized Controlled Prospective Study
Brief Title: Transversus Thoracic Plane Block for Perioperative Analgesia in Cardiac Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Joanna Tohme, Medical Doctor, Principal investigator, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEHDF2392
Record Dates: First submitted 2024-08-04; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Transversus Thoracic Plane Block; Cardiac Surgery; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (No Intervention): This group receives standard analgesic treatment and no Transversus Thoracic Plane Block is performed
- Transversus Thoracic Plane Block pre (Active Comparator): This group receives standard analgesic treatment and Transversus Thoracic Plane Block is performed before surgery
  Interventions: Procedure: Transversus Thoracic Plane Block
- Transversus Thoracic Plane Block post (Active Comparator): This group receives standard analgesic treatment and Transversus Thoracic Plane Block is performed at the end of surgery
  Interventions: Procedure: Transversus Thoracic Plane Block

INTERVENTIONS:
Procedure: Transversus Thoracic Plane Block — The Transversus Thoracic Plane Block is a recent regional anesthesia technique. It provides analgesia for the anterior cutaneous branches of the intercostal nerves T2-6 to the medial anterior chest wall via a single injection of local anesthesia between the internal intercostal muscle and the transversus thoracic muscle located between the third and fourth (or fourth and fifth) intercostal space. It is noteworthy that the TTPB can consequently reduce pulmonary morbidity and the need for high-dose opioids.
  Arms: Transversus Thoracic Plane Block post; Transversus Thoracic Plane Block pre

SUMMARY:
The goal of this clinical trial is to learn if perioperative Transversus Thoracic Plane Block (TTPB) decrease perioperative pain after cardiac surgery. The main questions it aims to answer are:

1. does Transversus Thoracic Plane Block decrease perioperative pain after cardiac surgery more than the standard analgesic treatment?
2. Are the results different if the investigators perform Transversus Thoracic Plane Block before surgery or at the end of surgery?

ELIGIBILITY:
Inclusion Criteria:

- All patients scheduled for cardiac surgery via sternotomy under cardiopulmonary bypass

Exclusion Criteria:

* Previous cardiac surgery
* Urgent surgery
* Pregnant women
* Allergy to local anesthetics
* Opioid dependence
* Low ejection fraction < 30%
* Presence or onset of cognitive or neurological disorders preventing pain assessment
* Infection at injection sites
* Coagulopathy
* Patients on dual antiplatelet therapy
* Renal insufficiency with Glomerular filtration rate (GFR) < 30 mL/min
* History of thoracic radiotherapy
* History of mastectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | First 24h postoperatively
  The primary outcome is Postoperative Pain Score:
  Numeric rating scale (NRS) ratings will be assessed at T1 (= upon patient awakening), T2 (= 12 hours postoperatively), T3 (= 24 hours postoperatively) as well as during various painful moments (coughing, drain removal, mobilization).
  Numeric rating scale (NRS) is a unidimensional measure of pain intensity. It consists of the patient evaluating his pain out of a series of numbers ranging from 0 to 10, where the 2 respective endpoints are "0 = no pain" and "10 = worst possible pain."

SECONDARY OUTCOMES:
Perioperative opioid requirement | First 24h postoperatively
  Total dose of opioids required during surgery and 24h postoperatively
Time to first opioid administration | First 24h postoperatively
  Time to first opioid administration after surgery
Time to extubation | First 24h postoperatively
  Time between arrival to cardiac intensive care unit and extubation
Patient satisfaction at 24 hours post surgery | First 24h postoperatively
  Patient satisfaction is measured by asking patients one question at 24 hours post surgery:
  "On a scale from 0 to 10, 0 = not satisfied at all, 10 = extremely satisfied, how satisfied do you feel concerning pain management during the first 24 hours after surgery? "
Length of stay at cardiac intensive care unit and hospital stay | 3 months postoperatively
  Length of stay at cardiac intensive care unit and hospital stay
Incidence of postoperative pneumonia and pneumothorax in cardiac intensive care unit | First 24h postoperatively
  Incidence of postoperative pneumonia and pneumothorax in cardiac intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Samia Madi Jebara, MD,PHD, Study Director — Saint-Joseph University
Locations (1):
- Hotel Dieu de France, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeanneteau A, Demarquette A, Blanchard-Daguet A, Fouquet O, Lasocki S, Riou J, Rineau E, Leger M. Effect of superficial and deep parasternal blocks on recovery after cardiac surgery: study protocol for a randomized controlled trial. Trials. 2023 Jul 6;24(1):444. doi: 10.1186/s13063-023-07446-2. PMID 37415221
- [Background] Wong HMK, Chen PY, Tang GCC, Chiu SLC, Mok LYH, Au SSW, Wong RHL. Deep Parasternal Intercostal Plane Block for Intraoperative Pain Control in Cardiac Surgical Patients for Sternotomy: A Prospective Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2024 Mar;38(3):683-690. doi: 10.1053/j.jvca.2023.11.038. Epub 2023 Nov 30. PMID 38148266
- [Background] Fujii S, Bairagi R, Roche M, Zhou JR. Transversus Thoracis Muscle Plane Block. Biomed Res Int. 2019 Jul 7;2019:1716365. doi: 10.1155/2019/1716365. eCollection 2019. PMID 31360703